CLINICAL TRIAL: NCT07367516
Title: A Phase Ib/II Clinical Trial Evaluating the Safety and Efficacy of TQB6411 Injection in Subjects With Recurrent or Metastatic Esophageal Cancer Who Have Failed Prior PD-1/PD-L1 Inhibitor Plus Platinum-Based Chemotherapy
Brief Title: Clinical Trial Evaluating TQB6411 Injection in Subjects With Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB6411-Ib/II-01
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB6411 Injection (Experimental): TQB6411 Injection , 21 days as a treatment cycle.
  Interventions: Drug: TQB6411 Injection

INTERVENTIONS:
Drug: TQB6411 Injection — TQB6411 Injection is an antibody-drug conjugate (ADC) targeting Epidermal Growth Factor Receptor (EGFR)/c-Met.

SUMMARY:
The Phase Ib stage of this study primarily aims to evaluate the tolerance and safety of TQB6411 Injection in subjects with recurrent or metastatic Esophageal cancer who have previously failed treatment with PD-1/PD-L1 monoclonal antibodies combined with platinum-based chemotherapy. The Phase II stage primarily aims to evaluate the efficacy of TQB6411 Injection in this same patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study, sign the informed consent form, and demonstrate good compliance.
* Age between 18 and 75 years old (inclusive)
* Eastern Cooperative Oncology Group (ECOG) score of 0-1
* Expected survival >12 weeks
* At least one measurable lesion per RECIST v1.1
* Laboratory criteria(no hematopoietic growth factor correction within 7 days)：

  * Hemoglobin (HGB) ≥90 g/L;
  * Absolute neutrophil count (NEUT) ≥1.5×10⁹/L;
  * Platelets (PLT) ≥90×10⁹/L;
  * Total bilirubin (TBIL) ≤1.5×ULN;
  * Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×ULN (≤5×ULN if liver metastases present);
  * Serum creatinine (CR) ≤1.3×ULNorcreatinine clearance rate (CCR) ≥50 mL/min;
* Histologically/cytologically confirmed recurrent or metastatic Esophageal cancer
* Failure/intolerance to prior PD-1/PD-L1 inhibitor plus platinum-based chemotherapy for recurrent/metastatic Esophageal Carcinoma (EC)
* Willingness to provide archived or fresh tumor tissue for biomarker analysis.
* Females of childbearing potential: Negative serum/urine pregnancy test within 7 days before enrollment and agreement to use effective contraception during and for 6 months post-study. Males: Agreement to use effective contraception during and for 6 months post-study.

Exclusion Criteria:

* Current or History of Other Malignancies
* Subjects with any condition that may compromise venous access for drug administration or blood sampling are excluded.
* Subjects with prior treatment-related adverse reactions that have not recovered to ≤ Grade 1 per CTCAE v5.0 criteria.
* Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose, Scheduled major surgery during the study intervention period, Non-healing wound, ulcer, or bone fracture at screening
* Subjects with any bleeding/hemorrhagic event ≥ Grade 3 (per CTCAE v5.0) occurring within 4 weeks before the first dose are excluded
* History of Thromboembolic Events within 6 Months
* Poorly Controlled Active Viral Hepatitis
* Subjects with active syphilis infection requiring antimicrobial therapy are excluded
* Subjects with any of the following pulmonary conditions are excluded: active tuberculosis, idiopathic pulmonary fibrosis (IPF), organizing pneumonia, drug-induced/radiation pneumonitis requiring treatment, symptomatic active pneumonia, or history of interstitial lung disease (ILD) requiring therapy
* History of Substance Abuse or Psychiatric Disorders
* History of Allogeneic Transplantation (Bone Marrow or Solid Organ)
* History of Hepatic Encephalopathy
* Major Cardiovascular Diseases
* Active or Uncontrolled Severe Infections
* Renal Failure Requiring Dialysis (Hemodialysis/Peritoneal Dialysis)
* History of Immunodeficiency
* Poorly Controlled Autoimmune Disease
* Poorly Controlled Autoimmune Disease & Epilepsy Requiring Treatment
* Poorly Controlled Diabetes
* Tumor-Related Symptoms and Treatment Considerations：

  * Exclusion Criterion - Recent Anticancer Treatment (≤3 Weeks or Within 5 Half-Lives)
  * Recent Use of National Medical Products Administration (NMPA) -Approved Anticancer Traditional Chinese Medicine (≤1 Week Prior to Treatment)
  * Radiologically Confirmed Tumor Encasement of Major Vessels with High Bleeding Risk
  * Uncontrolled Effusions Requiring Repeated Drainage
  * Known to have spinal cord compression, leptomeningeal metastasis/carcinomatous meningitis, or symptomatic brain metastases with less than 4 weeks of symptom/imaging control.
* Known Hypersensitivity to Investigational Drug or Excipients
* Prior Treatment with Topoisomerase I Inhibitor-Based ADCs and/or Irinotecan Chemotherapy
* Prior Participation in Anticancer Clinical Trials Within 4 Weeks
* Investigator-Assessed Safety or Compliance Concerns

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 3 mouths
  The RP2D is defined as the recommended dose for subsequent Phase II studies, which will be determined based on a comprehensive assessment of Pharmacokinetics (PK), preliminary efficacy, and safety.
Incidence and severity of adverse events | 24 mouths
  This study requires the collection of any adverse medical events occurring from the time the subject signs the informed consent form until 30 days after the last dose of study medication or the initiation of new anti-tumor therapy, whichever comes first.
Progression-Free Survival (PFS) | 24 mouths
  PFS is defined as the time from the first administration of treatment to the first occurrence of disease progression or death from any cause, whichever comes first, as determined by the investigator according to RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 mouths
  Proportion of patients with objective response(achieving Complete Response (CR) + Partial Response (PR) out of the total number of cases and 95% Confidence Interval (CI).
Disease Control Rate(Disease Control Rate=achieving Complete Response [CR] or+Partial Response [PR]+Stable Disease (SD) | 24 mouths
  Proportion of patients with disease control (achieving Complete Response [CR] or+Partial Response [PR]+Stable Disease[SD] out of the total number of cases and 95% CI.
Duration of Response (DOR) | 24 mouths
  DOR refers to the time interval from the first documentation of disease remission (achieving Complete Response [CR] or Partial Response [PR]) to the time of disease relapse or progression (PD).
Overall Survival (OS) | 24 mouths
  Overall Survival (OS) refers to the length of time from the date of diagnosis or the start of treatment for a disease (such as cancer) until the patient's death from any cause.
Peak plasma concentration (Cmax) | Within 14 days after administration
  It refers to the highest blood drug concentration achieved after administration of TQB6411 injection.
Area Under the Concentration-time Curve (AUC0-t) | Within 14 days after administration
  Area under the drug concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) after a single dose.
Area Under the Concentration-time Curve (AUC0-∞) | Within 14 days after administration
  Area under the drug concentration-time curve from time 0 extrapolated to infinity (AUC0-∞)
Peak time (Tmax) | Within 14 days after administration
  It refers to the time when the maximum blood drug concentration is reached after administration of TQB6411 for injection.
Number of subjects with incidence of anti-drug antibodies (ADA) and neutralizing antibodies (NAb) | 24 months
  Number and proportion of subjects positive for anti-drug antibodies (ADA) after treatment, along with 95% confidence intervals, and a description of the time of onset, titer, etc., of anti-drug antibody (ADA) development.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Tumor Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guangxi, Guizhou
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The Second People's Hosital of Jiaozuo, Jiaozuo, Henan
  - Luoyang Central Hospital (Zhengzhou University Affiliated Luoyang Central Hospital), Luoyang, Henan
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The first hospital of jilin university, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - Linyi cancer Hospital, Liyi, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi
  - Sichuan cancer hosipital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Zhongshan Hospital Fudan University, Shanghai